CLINICAL TRIAL: NCT01175122
Title: Phase 1 Evaluation of the Safety and Immunogenicity of Live Influenza A Vaccine H2N3 (6-2) AA ca Recombinant (A/Swine/Missouri/4296424/2006 (H2N3) x A/Ann Arbor/6/60 ca), a Live Attenuated Virus Vaccine Candidate for Prevention of Influenza H2N3 Infection in the Event of a Pandemic
Brief Title: Evaluation of the Safety and Immunogenicity of a Live Attenuated Virus Vaccine for the Prevention of H2N3 Influenza
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: URMC 10-004
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Influenza A Virus Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- H2N3 MO 2003/AA ca Vaccine (Experimental): Participants will receive a nasal spray administration of the H2N3 MO 2003/AA ca vaccine on Day 0 and Day 28.
  Interventions: Biological: H2N3 MO 2003/AA ca Vaccine

INTERVENTIONS:
Biological: H2N3 MO 2003/AA ca Vaccine — 0.2 mL of H2N3 MO 2003/AA ca vaccine delivered by an Accuspray nasal spray device on Day 0 and Day 28

SUMMARY:
In recent years, influenza viruses that have traditionally infected animals have infected humans as well. The H2N3 influenza virus, which first appeared in pigs in the Midwest United States in 2006, may pose a potential health concern to humans. This study will evaluate the safety of and immune response to a vaccine designed to protect people from the H2N3 influenza virus.

DETAILED DESCRIPTION:
Animal influenza viruses, such as the H1N1 and H5N1 viruses, typically infect animals like birds or pigs, but these viruses can also infect humans. The recent outbreak of the H1N1 influenza virus demonstrates that it is possible for these viruses to cause a pandemic outbreak in humans. Researchers are specifically interested in evaluating vaccines for H2 viruses, as these viruses caused a pandemic outbreak in humans in the late 1950s to 1960s. In addition, over half of the world's current population has no previous exposure to related viruses, which means a pandemic outbreak could pose a serious health risk as many people would have no immunity against the virus. In 2006, an outbreak of H2N3 infection occurred in pigs in the Midwest United States. While no humans contracted the virus during that outbreak, it remains a concern for researchers in the event that the virus ever spreads to humans. The purpose of this study is to evaluate the safety and immunogenicity of two doses of an experimental H2N3 vaccine, H2N3 MO 2006/AA ca in healthy adults. This is a live attenuated vaccine, which means that participants will be exposed to small amounts of the H2N3 vaccine virus and will need to remain isolated for at least 12 days when receiving the vaccine to prevent spreading the virus to others.

This study will enroll healthy adults. Participants will receive two doses of the vaccine, 4 weeks apart, and will stay in an isolation facility during both 12-day vaccination periods. Participants will be admitted to the isolation facility 2 days before they receive their first vaccination. They will receive one nasal spray administration of the vaccine and will be monitored for side effects. On various days while in the isolation facility, they will undergo a physical exam, blood and urine collection, and a nasal wash procedure. Participants will remain in the isolation facility for at least 9 days after receiving the vaccine and possibly longer, until the nasal wash tests negative for the vaccine virus for 2 consecutive days. Participants will be readmitted to the isolation facility 26 days after the first vaccination. They will receive a second vaccination and all study procedures will be repeated. Participants will attend study visits 56, 82, and 208 days after the first vaccination for follow-up health and safety monitoring, blood collection, and a nasal wash procedure.

ELIGIBILITY:
Inclusion Criteria:

* In general good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator
* Agree to storage of blood specimens for future research
* Available for the duration of the trial
* Willing to participate in the study as evidenced by signing the informed consent document
* Female participants must agree to use effective birth control methods for the duration of the study. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Pregnant or breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urine testing. Clinically significant alanine aminotransferase (ALT) levels, as determined by the principal investigator (PI), will be exclusionary at baseline, prior to vaccination.
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study procedures
* Previous enrollment in an H2 influenza vaccine trial or in any study of an avian influenza vaccine
* Seropositive to the H2N3 influenza A virus (serum HAI titer greater than 1:8)
* Positive urine drug toxicology test indicating narcotic use/dependency
* Have medical, occupational, or family problems as a result of alcohol or illicit drug use during the 12 months prior to study entry
* Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a person participating in the trial or would render the person unable to comply with the study procedures
* History of anaphylaxis
* Allergy to oseltamivir as determined by participant report
* Current diagnosis of asthma or reactive airway disease (within the 2 years prior to study entry)
* History of Guillain-Barré Syndrome
* Positive ELISA and confirmatory Western blot tests for human immunodeficiency virus-1 (HIV-1)
* Positive ELISA and confirmatory test (e.g., recombinant immunoblot assay) for hepatitis C virus (HCV)
* Positive hepatitis B virus surface antigen (HBsAg) by ELISA
* Known immunodeficiency syndrome
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to vaccination
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination
* History of a surgical splenectomy
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination
* Current smoker unwilling to stop smoking for the duration of the study. More information on this criterion can be found in the protocol.
* Travel to the Southern Hemisphere within 14 days prior to study vaccination
* Travel on a cruise ship within 14 days prior to study vaccination
* Receipt of another investigational vaccine or drug within 30 days prior to study vaccination
* Allergy to eggs or egg products

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events that occur during the acute monitoring (inpatient) phase of the study | Measured through Day 37 or until participants are discharged from the isolation unit
Area under the curve (AUC) of nasal virus shedding after each dose of vaccine as assessed by liquid titration of nasal secretions on Madin Darby canine kidney (MDCK) cells at 33°C | Measured after each vaccination
Development of serum antibody assessed by either hemagglutination inhibition (HAI) or microneutralization (MN) assays | Measured after each vaccination

SECONDARY OUTCOMES:
Development of a significant increase in nasal secretion hemagglutinin (HA)-specific antibody assessed by enzyme-linked immunosorbent assay (ELISA) | Measured until participants are discharged from the isolation unit
Development of greater than 200 influenza-specific interferon-gamma-secreting cells per million lymphocytes as assessed by enzyme-linked immuno spot assay (ELISPOT) on Day 28 after immunization | Measured 28 days after vaccination
Detection of influenza-specific IgG or IgA secreting B cells on Day 7 following vaccination assessed by antibody secreting cells (ASC) assay | Measured 7 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: John Treanor, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Background] Ma W, Vincent AL, Gramer MR, Brockwell CB, Lager KM, Janke BH, Gauger PC, Patnayak DP, Webby RJ, Richt JA. Identification of H2N3 influenza A viruses from swine in the United States. Proc Natl Acad Sci U S A. 2007 Dec 26;104(52):20949-54. doi: 10.1073/pnas.0710286104. Epub 2007 Dec 18. PMID 18093945
- [Background] Chen GL, Lamirande EW, Yang CF, Jin H, Kemble G, Subbarao K. Evaluation of replication and cross-reactive antibody responses of H2 subtype influenza viruses in mice and ferrets. J Virol. 2010 Aug;84(15):7695-702. doi: 10.1128/JVI.00511-10. Epub 2010 May 26. PMID 20504935